CLINICAL TRIAL: NCT06297512
Title: Interventional, Single-arm, Open-label Open-label, Phase II Trial to Evaluate the Role of Anthracycline Infusion After Radio Therapy (RT) in Pediatric and Young Adults With Glioblastoma (pGBM).
Brief Title: Evaluate the Role of Anthracycline After Radio Therapy in Patients With Glioblastoma (pGBM).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iacopo Sardi (Other)
Responsible Party: Sponsor-Investigator, Iacopo Sardi, Princiapl Investigator, Meyer Children's Hospital IRCCS
Organization: Meyer Children's Hospital IRCCS (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pGBM-WBRT/DOX2020
Record Dates: First submitted 2024-02-20; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pGBM patients therapy (Experimental): * Whole therapy radiation therapy
  * Temozolomide concomitant
  * After 1 month adjuvant Temozolomide,
  * After 3 months Doxorubicine
  * adjuvant Temozolomide
  Interventions: Drug: Radiotherapy, Temozolomide, Doxorubicin

INTERVENTIONS:
Drug: Radiotherapy, Temozolomide, Doxorubicin — Radiation treatment Concomitant TMZ: 75mg/m2/day per OS for 7 days per week, from the first day of radiotherapy to the last (maximum cumulative dose 3150mg/m2), with possibility of earlier initiation on clinician's judgment.
  After 1 month (4-5 weeks ± 7 days) from the end of RT/TMZ treatment they will receive:
  Adjuvant TMZ: 2 cycles at increasing doses (150-180 mg/m2) per OS for 5 consecutive days 28 days apart
  After 3 months (12 weeks ± 7 days) from the end of RT/TMZ treatment they will receive:
  Dox 4 cycles with 37.5mg/m2/day by continuous infusion over 48 hours (2 days) every 28 days (maximum cumulative dose 300mg/m2)
  And after 4 weeks ± 7 days from the end of Dox treatment they will receive:
  TMZ adjuvant 12 cycles at increasing doses (150-180 mg/m2) by OS for 5 consecutive days 28 days apart (maximum cumulative dose 16200 mg/m2);

SUMMARY:
Glioblastoma (GBM) and diffuse intrinsic bridge gliomas (DIPG) only the most aggressive forms of cancer, and their prognosis remains bleak. Currently, the standard of treatment is TMZ concomitant with radiotherapy, and, at the end of combined treatment, as adjuvant therapy. In vitro and in vivo experimental studies have suggested that anthracyclines are effective antineoplastics for the treatment of gliomas. In patients with solid tumors treated with anthracyclines, continuous infusion administration compared with bolus administration has been shown to provide a better safety profile especially with regard to cardiotoxicity. Based on this evidence, this study aims to evaluate the safety and antitumor activity of combined treatment with Dox, WBRT (whole body radiotherapy), and TMZ in pediatric and young adult patients affected by GMB

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological-molecular diagnosis according to WHO 2016 classification: IDH-wildtype glioblastoma (9440/3), giant cell glioblastoma (9441/3), gliosarcoma (9442/3), epithelioid glioblastoma (9440/3), IDH-mutated glioblastoma (9445/3), glioblastoma NOS (9440/3), diffuse astrocytoma (9400/3), diffuse midline glioma H3 K27M mutated, including multifocal, metastatic or gliomatosis cerebri pictures of first diagnosis Not previously treated (with chemo and radiotherapy) or treated only surgically (total, near partial, partial, biopsy).
* Males and females between the ages of 3 and 30 years old
* Life expectancy ≥ 12 months
* karnofsky/Lansky ≥ 80 %
* Adequate hematologic function: Absolute leukocyte count ≥ 2.0 x 109/l, Hemoglobin ≥ 10 g/dl, Platelet count ≥ 50 x 109/l
* Adequate liver function: Total bilirubin ≤ 2.5 x ULN, ALT/AST ≤ 5.0 x ULN
* Adequate renal function:Serum creatinine ≤ 1.5 x ULN
* Written informed consent from the patient, parents or legal guardians
* Patient's willingness during treatment and ability to comply with the protocol

Exclusion Criteria:

* Evidence of any other serious disease or condition that is a contraindication to study therapy (e.g. severe mental retardation, severe cerebral palsy, severe syndromes congenital syndromes, heart disease)
* Performance of a course of 1st-line chemotherapy at the same time as study initiation
* Concurrent participation in other research projects
* Pregnancy or lactation status
* Use of inappropriate contraceptive methods

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2027-11-09 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation prolonged Dox | through study completion, an average of 1 year
  Time to early withdrawal from experimental treatment with Dox
Percentage of Withdrawal from the study rate | through study completion, an average of 1 year
  Percentage of subjects with SAE leading to withdrawal from the study
Percentage of SAEs | through study completion, an average of 1 year
  Percentage of SAEs
Mortality rate | through study completion, an average of 1 year
  Mortality from adverse events
Early discontinuation of dox treatment rate | through study completion, an average of 1 year
  Proportion of early discontinuation of experimental treatment with Dox

SECONDARY OUTCOMES:
Event-free survival (EFS), disease progression (PFS), and overall survival (OS) | through study completion, an average of 1 year
  Event-free survival (EFS) calculated as the time between the date of enrolment and the date of occurrence of one of the events:
  * disease progression established according to the modified RANO criteria for paediatric age
  * clear progression of non-measurable lesions (T1);
  * - any new lesion;
  * clinical deterioration due to the tumour and not attributable to other causes (e.g, seizures, adverse drug effects, complications of therapy, cerebrovascular events infections and so on);
  * failure to return for evaluation following death (from any cause) or deterioration of condition;
  * and other described in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Iacopo Sardi, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy